CLINICAL TRIAL: NCT02652832
Title: Effects of Noninvasive Brain Stimulation Techniques on BDNF Levels
Acronym: Plasti-Stim
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: CSR B04
Record Dates: First submitted 2015-10-19; First posted 2016-01-12 (Estimated); Last update posted 2018-08-01 (Actual); Status verified 2018-02

CONDITIONS: Depression; Schizophrenia
MeSH Terms: conditions — Depression; Schizophrenia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Depression Electroconvulsive therapy (Active Comparator): 40 patients with major depression receiving a mean of 12 sessions of Electroconvulsive therapy
  Interventions: Device: non invasive brain stimulation
- Depression active repetitive transcranial magnetic stimulation (Active Comparator): 40 patients with major depression receiving a mean 4 weeks of 1 Hz repetitive transcranial magnetic stimulation applied over the right dorsolateral prefrontal cortex - DLPFC
  Interventions: Device: non invasive brain stimulation
- Depression sham repetitive transcranial magnetic stimulation (Sham Comparator): 40 patients with major depression receiving a mean 4 weeks of sham 1 Hz repetitive transcranial magnetic stimulation applied over the right dorsolateral prefrontal cortex - DLPFC
  Interventions: Device: non invasive brain stimulation
- Schizophrenia active transcranial magnetic stimulati (Active Comparator): 40 patients with schizophrenia and predominant negative symptoms receiving 20 sessions of intermittent theta burst simulation (iTBS) applied over the left dorsolateral prefrontal cortex - DLPFC
  Interventions: Device: non invasive brain stimulation
- Schizophrenia sham transcranial magnetic stimulation (Sham Comparator): patients with schizophrenia and predominant negative symptoms receiving 20 sessions of sham intermittent theta burst simulation (iTBS) applied over the left dorsolateral prefrontal cortex - DLPFC
  Interventions: Device: non invasive brain stimulation
- Schizophrenia active transcranial Direct Current Stimulation (Active Comparator): 40 patients with schizophrenia and auditory verbal hallucinations receiving 10 sessions of transcranial Direct current stimulation (tDCS) applied with the anode over the left dorsolateral prefrontal cortex - DLPFC- and the cathode over the left temporoparietal junction
  Interventions: Device: non invasive brain stimulation
- Schizophrenia sham transcranial Direct Current Stimulation (Sham Comparator): 40 patients with schizophrenia and auditory verbal hallucinations receiving 10 sessions of sham transcranial Direct current stimulation (tDCS) applied with the anode over the left dorsolateral prefrontal cortex - DLPFC- and the cathode over the left temporoparietal junction
  Interventions: Device: non invasive brain stimulation
- Healthy volunteers (No Intervention): 80 healthy volunteers receiving no stimulation

INTERVENTIONS:
Device: non invasive brain stimulation — non invasive brain stimulation
  Other Names: rTMS; tDCS; ECT
  Arms: Depression Electroconvulsive therapy; Depression active repetitive transcranial magnetic stimulation; Depression sham repetitive transcranial magnetic stimulation; Schizophrenia active transcranial Direct Current Stimulation; Schizophrenia active transcranial magnetic stimulati; Schizophrenia sham transcranial Direct Current Stimulation; Schizophrenia sham transcranial magnetic stimulation

SUMMARY:
The aim of this study is to investigate the effects of non invasive brain stimulation - NIBS - techniques (Electroconvulsivotherapy - ECT, transcranial Direct Current Stimulation - tDCS, repetitive transcranial magnetic stimulation - rTMS) on serum Brain Derived Neurotrophic factor (BDNF) levels in patients with depression and schizophrenia. Four blood samples will be collected in each participants, one before the NIBS sessions, and 3 after the completion of NIBS protocols: one immediately after the end of the NIBS sessions, a second one week after and a last one month after. Two blood samples separated by one month will also be collected in a a group of healthy volunteers.

DETAILED DESCRIPTION:
The hypothesis is that NIBS will modulate BDNF levels and that the modification in serum BDNF levels will be correlated with clinical improvements in the sample of patients.

ELIGIBILITY:
Inclusion Criteria:

* in the depression group: DSM IV criteria of MDD; HDRS17> 22; stage 2 of resistance; received rTMS or ECT
* in the schizophrenia group DSM IV criteria of schizophrenia; pharmaco-resistance of symptoms (either negative symptoms or auditory verbal hallucination); received rTMS or tDCS
* in the healthy volunteers group : to not have axis I of DSM IV diagnosis; no siblings with axis I DSM IV diagnosis

Exclusion Criteria:

* less than 18 years old
* pregnancy
* received benzodiazepine

In the depression and schizophrenia group:

* bipolar disorder
* other axis I of DSM IV diagnosis (excluding for Tobacco use disorder)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2010-12 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
serum BDNF levels | from baseline to one month

CONTACTS AND LOCATIONS:
Overall Officials: jerome brunelin, PhD, Study Director — CH le vinatier
Locations (1):
- Hopital Le vinatier, Bron, France